CLINICAL TRIAL: NCT07175181
Title: Impact of Gut Microbiota on Clinical Outcomes and Left Ventricular Remodeling After Primary Percutaneous Coronary Intervention
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Gamal AbdelHakam, Residant doctor at Assiut university hospital, Assiut University
Other Study IDs: Microbiota PCI
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Primary Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A: patients Confirmed diagnosis of ST-elevation myocardial infarction (STEMI) and indication for PCI based on clinical guidelines

SUMMARY:
Left ventricular remodeling (LVR) refers to the structural and functional changes that occur in the left ventricle following myocardial injury. These changes can include alterations in left ventricular shape, size, wall thickness, and volume, which can ultimately lead to decreased cardiac function and increased risk of heart failure. The remodeling process is often maladaptive and can worsen the prognosis of patients with CAD. Recent advances in microbiome research have unveiled the critical role of gut microbiota in modulating systemic health, including cardiovascular health. The gut microbiome consists of trillions of microorganisms that engage in complex interactions with the host, influencing various physiological processes. Among these interactions is the production of metabolites that can directly affect cardiovascular physiology. Notably, Trimethylamine N-oxide (TMAO). Elevated TMAO levels have been associated with increased risk of atherosclerosis and cardiovascular events, including those following PCI. Data suggest that TMAO may promote endothelial dysfunction and enhance inflammatory pathways, thereby exacerbating vascular injury and LV remodeling. These findings indicate that the interaction between gut microbiota composition, TMAO production, and cardiovascular risk could represent a novel therapeutic target for improving patient outcomes after PCI . Understanding the dynamics of these relationships can provide critical insights into individualized treatment strategies and dietary interventions that may mitigate cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years .
* Confirmed diagnosis of ST-elevation myocardial infarction (STEMI) and indication for PCI based on clinical guidelines.
* Patients scheduled to undergo primary PCI for STEMI.
* Ability and willingness to provide informed consent for participation and for the collection of stool samples.
* No significant comorbidities that may confound the results (e.g., chronic kidney disease, liver cirrhosis).
* No prior use of antibiotics, probiotics, or prebiotics within the last 3 months, as these may significantly alter gut microbiota composition.
* Willingness and ability to complete follow-up assessments as required by the study protocol.
* Absence of major gastrointestinal disorders (e.g., inflammatory bowel disease, gastrointestinal infections) that could affect gut microbiota.

Exclusion Criteria:

* Age < 18 years.
* Chronic Diseases:

  * Chronic kidney disease (stage 3 or higher).
  * Chronic liver disease (e.g., cirrhosis).
  * Active malignancies.
* Acute infections or active inflammatory conditions at the time of PCI.
* Gastrointestinal Disorders:

  * Inflammatory bowel disease.
  * Celiac disease.
  * Diverticulitis.
* Recent use of antibiotics, probiotics, or prebiotics within the last 3 months.
* Use of immunosuppressive medications or chemotherapy.
* Uncontrolled diabetes or hypertension.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Confirmed diagnosis of ST-elevation myocardial infarction (STEMI) and indication for PCI based on clinical guidelines.
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Plasma levels of Trimethylamine N-oxide (TMAO) | baseline
  Measurement: Plasma levels of Trimethylamine N-oxide (TMAO) will be quantified before or after PCI, using ELISA kits or other validated methods.